CLINICAL TRIAL: NCT00754026
Title: Influence of the Insertion Distance on Loss of Sensation Produced by Interscalene Perineural Catheters in the Context of Shoulder Surgery.
Brief Title: Insertion Distance of Interscalene Perineural Catheters in the Context of Shoulder Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Dr Geneviève Arcand, Centre Hospitalier de l'Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08.072
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Pain
Keywords: Shoulder surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Procedure: Insertion of interscalene catheter for shoulder surgery
- 2 (Active Comparator)
  Interventions: Procedure: Insertion of interscalene catheter for shoulder surgery

INTERVENTIONS:
Procedure: Insertion of interscalene catheter for shoulder surgery — Distance of interscalene catheter: 2cm
  Arms: 1
Procedure: Insertion of interscalene catheter for shoulder surgery — Distance of interscalene catheter: 6cm
  Arms: 2

SUMMARY:
This study is designed to compare interscalene catheter insertion distances, in order to determine which is the best for pain relief after shoulder surgery.

DETAILED DESCRIPTION:
Pain following shoulder surgery is reported as severe for 70% of patients, and is a major concern in both hospitalised and ambulatory surgery patients. Pain control is particularly important, as adequate analgesia allows rapid mobilisation of the operated shoulder and prevents complications related to immobility. Several methods have been proposed to treat this pain, the most promising being the interscalene nerve block. The injection of local anesthetics reduces sensation from the shoulder and provides better pain relief after surgery than narcotic medication. To prolong the duration of the analgesia, a catheter must be positioned next to the brachial plexus. Through this catheter, small quantities of local anesthetics can be continuously delivered for several hours after surgery, effectively relieving the worst of the pain.

To date, the continuous interscalene nerve block has been shown to improve pain relief, to reduce nausea, vomiting, pruritus and sleep disturbances after shoulder surgery. It also reduces the need for opioids.

Until recently, catheter techniques were not frequently used due to technical difficulties encountered with catheter installation and catheter displacement after surgery. Due to recent improvements in nerve and catheter localisation, catheter installation has become easier, more precise and more reliable. However, the distance at which the catheter must be advanced next to the brachial plexus in order to provide the best pain relief remains unknown. Insertion distance could influence the initial quality and distribution of the freezing, its duration, or both. Therefore, this study is designed to compare two catheter insertion distances, in order to help determine which is best for pain relief after shoulder surgery.

Methods :

1. Insertion of the catheter :

   Patients will be randomly assigned to the following groups :
   * Group 1 : 2 cm insertion
   * Group 2 : 6 cm insertion

   The anesthesiologist will insert the interscalene catheter before the beginning of anesthesia for surgery. The usual medication will be used to make the installation of the catheter comfortable. Standard non-invasive monitoring will be used. The exact location where the catheter will be put in place will be identified using an ultrasound machine. This device will allow the anesthesiologist to identify the various anatomical structures. A specially designed needle will be inserted next to the brachial plexus and its position will be confirmed with a neurostimulator. Once the adequacy of needle position is confirmed, the anesthesiologist will introduce 2 cm (Group 1) or 6 cm (Group 2) of the catheter through the needle, and then will withdraw the needle. The catheter will be fixed in place to avoid displacement.

   Patients will receive standard regional or general anesthesia for this type of surgery.
2. Post-operative analgesia :

   * All patients : patients will receive, through the interscalene catheter, a continuous infusion of bupivacaine 0,15% at the rate of 5 mL/h for at least 24 hours post-operatively After surgery, pain will be assessed using a verbal numeric pain scale. Patients will be asked to fill out a pain intensity measurement form using a 0-10 pain scale at 3, 6 and 24 hours after surgery.
   * Inpatients : along with the infusion; a Patient Controlled Analgesia pump will be provided to the patients.
   * Ambulatory patients : the infusion will be given through a disposable elastomeric pump. Along with the infusion, patients will receive oral hydromorphone to complete pain relief. Patients will receive standard post-operative instructions on the use of the pump and catheter. Telephone and pager numbers for physicians available at all time will also be provided to each patient. They will be asked to record their opioid use on a medication log for the first 24 hours post-operatively.

   Sensory block will be assessed in the major nerve distributions of the arm at 24 h after surgery. Ambulatory patients will be invited to return to the hospital to have this assessment performed.
3. Follow-up

All patients will receive a phone call from the research team one week after surgery to assess their satisfaction towards the analgesia and to inquire about potential complications of the interscalene block.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older undergoing elective shoulder surgery

Exclusion Criteria:

* Severe COPD
* Coagulopathy
* Allergy to local anesthetics
* Chronic use of opioids
* Peripheral neuropathy of the operated limb
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Sensory block assessment | 24 hours after surgery

SECONDARY OUTCOMES:
Quality of pain relief | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève Arcand, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (Hôpital Notre-Dame), Montreal, Quebec, Canada